CLINICAL TRIAL: NCT02817269
Title: Referred Pain Patterns in Trigger Point 2 of the Infraspinatus Muscle in Patients With Shoulder Pain
Brief Title: Referred Pain Patterns Infraspinatus Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Emilio-José Poveda-Pagán, PhD, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: UniversidadMHE-1
Record Dates: First submitted 2016-06-21; First posted 2016-06-29 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Shoulder Pain
Keywords: Shoulder pain; Trigger points; Referred pain; Visual analogue scale
MeSH Terms: conditions — Shoulder Pain; Pain, Referred

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual palpation group (Experimental): For the manual palpation group, the reference position will be a lateral position, lying on the non affected shoulder while the affected side will be explored. The arm and elbow are flexed 90° resting on a pillow and legs placed with 90° hip and knee flexion to stabilize the body, with the head resting on a pillow to maintain body alignment. The physiotherapist will be in front of the participant and carried out the examination with flat palpation using the thumb to identify soreness taut band tried to elicit local twitch response and referred pain in the infraspinatus area. First, three attempts will be made to elicit an local twitch response (LTR) using snapping palpation if a response will be obtained. After LRT, referred pain could also be evoked by palpation.
  Interventions: Other: Manual palpation
- Deep dry needling group (Experimental): For the deep dry needling group, the reference position will be a lateral position, lying on the non affected shoulder while the affected side will be explored. The arm and elbow are flexed 90° resting on a pillow and legs placed with 90° hip and knee flexion to stabilize the body, with the head resting on a pillow to maintain body alignment. The physiotherapist will be in front of the participant and carried out the examination with flat palpation using the thumb to identify soreness taut before making the needle insertion. Sterile stainless steel needles (length 40mm/caliber 0.32 with a cylindrical plastic guide) will be used.
  Interventions: Other: Deep dry needling

INTERVENTIONS:
Other: Manual palpation — The manual palpation level will kept constant by applying enough digital pressure to cause the finger nail bed to blanch. When the nail will be turn pale, the amount of pressure will be measured at approximately 3 4kg/cm2 and will be maintained for 5-10 seconds to evoke referred pain. A manual palpation referred pain will be present if the pain radiated far enough for the patient to feel more than just a local pain.
  Arms: Manual palpation group
Other: Deep dry needling — Intramuscular needling will be carried out via deep dry needling into myofascial trigger point (MTrP) area without the introduction any substances. The aim is to elicit a local twitch response upon inserting the needle into the MTrP area and perform a neurological stimulation (by rotating the needle 360 degrees) to more easily evoke referred pain, holding for 10 seconds and then extracting the needle gently. The procedure will be followed by one minute of haemostatic compression.
  Arms: Deep dry needling group

SUMMARY:
The first aim of the study will be to identify the most common ReP pattern and compare its coincidence with that described by Travell and Simons. Second, the study aim will be to verify whether there are any significant differences by sex and types of technique used in regard to the ReP pattern of TrP 2 of the infraspinatus muscle, an area described as more sensitive.Finally, the third aim of the study will be to determine whether deep dry needling will evoke the LTR and ReP more easily than manual palpation.

DETAILED DESCRIPTION:
Patients will be recruited from a university's employee and student population by advertising at the university. Patients with shoulder complaints (described as pain felt in the shoulder or upper arm) will be randomly assigned to either an manual palpation or deep dry needling group. Participants will be randomly divided into 2 groups, a deep dry needling group and manual palpation group. Visual analogue scale (VAS), referred pain (ReP) pattern and features of referred pain of the infraspinatus muscle will be all assessed post-technique.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years.
* To remain seated or in front of data visualization screens (tablets, computers or smartphones) for at least 4 hours a day.
* Shoulder complaints in the last six weeks.

Exclusion Criteria:

* Patients with evidence of serious medical illness.
* Cognitive impairment.
* Psychosocial disorders.
* Bilateral affectation of shoulder pain.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Mapping of Referred Pain Pattern | One month
  The participants from both groups will ask to report whether ReP is evoked and to describe the ReP pattern using an anatomical map of the upper half of the human body divided into eighteen areas. Nine areas corresponded to the anterior part of the body and the other nine to the posterior part of the body.

SECONDARY OUTCOMES:
Prevalence active trigger point | One month
  Active trigger point is considered: Soreness taut band and familiar pain.
Evocation of Local Twitch Response | One month
  These were assigned a numerical value of 0 (yes) or 1 (no) for better statistical handling of the data.
Subjective pain intensity: Visual Analogue Scale (VAS) | One month
  The VAS for pain measures the amount of pain experienced by a subject on a continuum from 0 to 10, with 0 being no pain and 10 maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: José V Segura-Heras, PhD in math, Study Chair — UNIVERSIDAD MIGUEL HERNÁNDEZ DE ELCHE (ALICANTE)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Audette JF, Wang F, Smith H. Bilateral activation of motor unit potentials with unilateral needle stimulation of active myofascial trigger points. Am J Phys Med Rehabil. 2004 May;83(5):368-74, quiz 375-7, 389. doi: 10.1097/01.phm.0000118037.61143.7c. PMID 15100626
- [Result] Borg-Stein J. Management of peripheral pain generators in fibromyalgia. Rheum Dis Clin North Am. 2002 May;28(2):305-17. doi: 10.1016/s0889-857x(02)00004-2. PMID 12122919
- [Result] Bron C, Dommerholt J, Stegenga B, Wensing M, Oostendorp RA. High prevalence of shoulder girdle muscles with myofascial trigger points in patients with shoulder pain. BMC Musculoskelet Disord. 2011 Jun 28;12:139. doi: 10.1186/1471-2474-12-139. PMID 21711512
- [Result] Bron C, Wensing M, Franssen JL, Oostendorp RA. Treatment of myofascial trigger points in common shoulder disorders by physical therapy: a randomized controlled trial [ISRCTN75722066]. BMC Musculoskelet Disord. 2007 Nov 5;8:107. doi: 10.1186/1471-2474-8-107. PMID 17983467
- [Result] Chou LW, Hsieh YL, Kuan TS, Hong CZ. Needling therapy for myofascial pain: recommended technique with multiple rapid needle insertion. Biomedicine (Taipei). 2014;4(2):13. doi: 10.7603/s40681-014-0013-2. Epub 2014 Aug 2. PMID 25520926
- [Result] Ge HY, Fernandez-de-Las-Penas C, Madeleine P, Arendt-Nielsen L. Topographical mapping and mechanical pain sensitivity of myofascial trigger points in the infraspinatus muscle. Eur J Pain. 2008 Oct;12(7):859-65. doi: 10.1016/j.ejpain.2007.12.005. Epub 2008 Jan 18. PMID 18203637